CLINICAL TRIAL: NCT06525961
Title: A Single-center, Open-label, Single-arm Study to Evaluate the Effectiveness and Safety of Extra Nasal Neurostimulator in Patients With Dry Eye Disease Dissatisfied With Artificial Tears
Brief Title: iTear Single-center, Open-label, Single-arm Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: ARCTIC VISION HONG KONG BIOTECH LIMITED (Unknown)
Responsible Party: Principal Investigator, Allie Lee, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: itear2024
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye Disease; Dry Eye Syndromes; Dry Eye; Meibomian Gland Dysfunction
Keywords: Dry Eye; DED; Dry Eye Syndromes; Meibomian Gland Dysfunction (MGD)
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Participants with iTEAR100 Neurostimulator (Experimental): The participants will use iTEAR100 Neurostimulator for the stimulation of the anterior ethmoidal nerve - which is located at the point between bony and fleshy tissue alongside the nose. Participants should apply stimulation to each side of the nose for 30 seconds, twice a day. It is recommended to apply once in the morning and once in the evening.
  Interventions: Device: iTEAR100 Neurostimulator

INTERVENTIONS:
Device: iTEAR100 Neurostimulator — To apply an iTEAR100 Neurostimulator for the stimulation to the anterior ethmoidal nerve - which is located at the point between bony and fleshy tissue alongside the nose. Participants should apply stimulation to each side of the nose for 30 seconds, twice a day. It is recommended to apply once in the morning and once in the evening.

SUMMARY:
This study aims to evaluate the effectiveness and safety of a device, iTEAR100 Neurostimulator (the device), which is designed to help people with Dry Eye Disease (DED) who are not satisfied with using artificial tears. The study will last three months and take place at one location. Thirty participants will use the iTEAR100 Neurostimulator, which stimulates the outside of the nose to help with dry eye symptoms.

Participants will have three main visits: one at the start (Day 0), one after 30 days (Day 30), and one at the end of the study (Day 90). For the first 30 days, they will use the device twice a day for 30 seconds on each side of the nose. After that, they will use it as needed for the next 60 days.

Before starting the treatment, participants will undergo tests to measure their initial eye condition. The effectiveness of the device will be checked by comparing these baseline measurements to those taken on Day 30 and Day 90. Participants will also fill out a questionnaire about their eye symptoms on Day 14.

The main measure of success is how much the participants' symptoms improve on the Ocular Surface Disease Index (OSDI) from Day 0 to Day 30. Other measures include changes in tear production, tear quality, and eye health from Day 0 to Days 30 and 90. Participants' safety will be monitored by tracking any adverse events (side effects) throughout the study.

DETAILED DESCRIPTION:
This is a Phase IV, single-centre, open-label, single-arm study to evaluate the effectiveness and safety of extra nasal neurostimulation in relieving symptoms of patients with Dry Eye Disease (DED) who are dissatisfied with artificial tear treatment. The intervention product is the extranasal neurostimulator, branded iTEAR.

The study duration is three months, with visits on Days 0, 30 and 90. Participants will follow a treatment regimen to apply neurostimulation to each side of the nose for 30 seconds twice daily for 30 days. From Day 31 to Day 90, participants will use the device as needed. Screening tests to measure baseline levels will be performed on Visit 1, and efficacy measures will be performed on Day 30 and Day 90. The participants will be instructed to perform a questionnaire on the ocular surface disease index (OSDI) on Day 14. Primary efficacy measures include changes in OSDI from baseline to Day 30. Secondary efficacy measures include the change in Schirmer Test Score, tear lipid layer thickness, corneal/conjunctival staining, and non-invasive tear film break-up time (NIBUT) from baseline to Day 30 and Day 90. Adverse Event (AE) Query is used as a safety measure to report adverse events in the duration of the study. The estimation of subjects in this trial is 30, with a power of 0.8 and assuming a 20% dropout rate.

To be included in the study, participants must be able to provide informed consent to participate in the study. They must have reported dissatisfaction (OSDI ≥ 23) with the recent use of artificial tears for DED (within 30 days of Visit 1), and Schirmer Test Score ≤ 10 mm/5 min in at least one eye.

The study eye will be defined as the eye with a Schirmer Test Score ≤ 10 mm/5 min. If both eyes qualify, the eye with a lower Schirmer Test Score during screening will be chosen as the study eye. If there is no difference, the right eye will be selected as the study eye.

The participants are excluded from the study if they have used extranasal or intranasal neurostimulator within 30 days of Visit 1, or participated in any clinical trial with an investigational substance or device within 30 days of Visit 1. In the opinion of the investigator, any condition that could impair study participation/ocular evaluation, or the potential risks of participation outweigh the potential benefits will also lead to exclusion from the study.

The participants will be withdrawn from the study if they voluntarily withdraw their consent to study participation, develop any adverse event that prevents the study participation, persistently do not comply with the study protocol, are lost to follow-up, or when the investigator believes the risk of further subject participation outweighs the benefit.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all the following criteria to be enrolled in this study:

1. Provided informed consent, approved by the Institutional Review Board (IRB), to participate in the study.
2. Reported use of artificial tears for DED within 30 days of Visit 1.
3. Ocular Surface Disease Index (OSDI) ≥ 23 (with no more than 3 N/A in the answers).
4. Anesthetized Schirmer Test Score ≤ 10 mm/5 min in at least one eye.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Used extranasal or intranasal neurostimulator within 30 days of Visit 1.
2. Participation in any clinical trial with an investigational drug or device within 30 days of Visit 1.
3. In the opinion of the investigator, any condition that could impair study participation/ocular evaluation or the potential risks of participation outweigh the potential benefits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
OSDI Score | 30 Days from baseline
  Change in OSDI at Day 30 from Baseline (Statistical testing using one-sided one-sample t-test)

SECONDARY OUTCOMES:
OSDI Score | Day 14 and Day 90 from baseline
  1. Change in OSDI from baseline to Day 14 and Day 90
Schirmer Test | Day 30 and Day 90 from baseline
  2. Change in Schirmer Test Score from baseline to Day 30 and Day 90
Lipid Layer Thickness (Pre) | Day 30 and Day 90 from baseline
  3. Change in tear lipid layer thickness (pre-stimulation) from baseline to Day 30 and Day 90
Lipid Layer Thickness (Pre vs Post) | Day 14, Day 30, Day 90
  4. Change between pre-stimulation and post-stimulation of tear lipid layer thickness in each visit
Corneal/Conjunctival Staining | Day 30 and Day 90 from baseline
  6. Change in Corneal/Conjunctival Staining from baseline to Day 30 and Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Allie LEE, Dr., Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Ophthalmology, LKS Faculty of Medicine, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Asbell PA, Maguire MG, Peskin E, Bunya VY, Kuklinski EJ; Dry Eye Assessment and Management (DREAM(c)) Study Research Group. Dry Eye Assessment and Management (DREAM(c)) Study: Study design and baseline characteristics. Contemp Clin Trials. 2018 Aug;71:70-79. doi: 10.1016/j.cct.2018.06.002. Epub 2018 Jun 6. PMID 29883769
- [Background] Asbell P, Vingrys AJ, Tan J, Ogundele A, Downie LE, Jerkins G, Shettle L. Clinical Outcomes of Fixed Versus As-Needed Use of Artificial Tears in Dry Eye Disease: A 6-Week, Observer-Masked Phase 4 Clinical Trial. Invest Ophthalmol Vis Sci. 2018 May 1;59(6):2275-2280. doi: 10.1167/iovs.17-23733. PMID 29715369
- [Background] Friedman NJ, Butron K, Robledo N, Loudin J, Baba SN, Chayet A. A nonrandomized, open-label study to evaluate the effect of nasal stimulation on tear production in subjects with dry eye disease. Clin Ophthalmol. 2016 May 4;10:795-804. doi: 10.2147/OPTH.S101716. eCollection 2016. PMID 27217719
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Dieckmann GM, Cox SM, Lopez MJ, Ozmen MC, Yavuz Saricay L, Bayrakutar BN, Binotti WW, Henry E, Nau J, Hamrah P. A Single Administration of OC-01 (Varenicline Solution) Nasal Spray Induces Short-Term Alterations in Conjunctival Goblet Cells in Patients with Dry Eye Disease. Ophthalmol Ther. 2022 Aug;11(4):1551-1561. doi: 10.1007/s40123-022-00530-x. Epub 2022 Jun 2. PMID 35653029
- [Background] Dieckmann, G., Kataguiri, P., Pondelis, N., Jamali, A., Alessandro Abbouda, salem, zeina, Franke, M., Senchyna, M., & Hamrah, P. (2017). In Vivo Confocal Microscopy Demonstrates Intranasal Neurostimulation-Induced Goblet Cell Alterations in Patients with Dry Eye Disease. Investigative Ophthalmology & Visual Science, 58(8), 2694-2694.
- [Background] Eom Y, Lee JS, Kang SY, Kim HM, Song JS. Correlation between quantitative measurements of tear film lipid layer thickness and meibomian gland loss in patients with obstructive meibomian gland dysfunction and normal controls. Am J Ophthalmol. 2013 Jun;155(6):1104-1110.e2. doi: 10.1016/j.ajo.2013.01.008. Epub 2013 Mar 7. PMID 23465270
- [Background] Gupta A, Heigle T, Pflugfelder SC. Nasolacrimal stimulation of aqueous tear production. Cornea. 1997 Nov;16(6):645-8. PMID 9395874
- [Background] Ji MH, Moshfeghi DM, Periman L, Kading D, Matossian C, Walman G, Markham S, Mu A, Jayaram A, Gertner M, Karpecki P, Friedman NJ. Novel Extranasal Tear Stimulation: Pivotal Study Results. Transl Vis Sci Technol. 2020 Nov 17;9(12):23. doi: 10.1167/tvst.9.12.23. eCollection 2020 Nov. PMID 33244443
- [Background] Kim J, Kim JY, Seo KY, Kim TI, Chin HS, Jung JW. Location and pattern of non-invasive keratographic tear film break-up according to dry eye disease subtypes. Acta Ophthalmol. 2019 Dec;97(8):e1089-e1097. doi: 10.1111/aos.14129. Epub 2019 May 6. PMID 31062499
- [Background] Gumus K, Schuetzle KL, Pflugfelder SC. Randomized Controlled Crossover Trial Comparing the Impact of Sham or Intranasal Tear Neurostimulation on Conjunctival Goblet Cell Degranulation. Am J Ophthalmol. 2017 May;177:159-168. doi: 10.1016/j.ajo.2017.03.002. Epub 2017 Mar 14. PMID 28302532
- [Background] Simmons PA, Liu H, Carlisle-Wilcox C, Vehige JG. Efficacy and safety of two new formulations of artificial tears in subjects with dry eye disease: a 3-month, multicenter, active-controlled, randomized trial. Clin Ophthalmol. 2015 Apr 15;9:665-75. doi: 10.2147/OPTH.S78184. eCollection 2015. PMID 25931807
- [Background] Verjee MA, Brissette AR, Starr CE. Dry Eye Disease: Early Recognition with Guidance on Management and Treatment for Primary Care Family Physicians. Ophthalmol Ther. 2020 Dec;9(4):877-888. doi: 10.1007/s40123-020-00308-z. Epub 2020 Oct 22. PMID 33090327
- [Background] Williamson JF, Huynh K, Weaver MA, Davis RM. Perceptions of dry eye disease management in current clinical practice. Eye Contact Lens. 2014 Mar;40(2):111-5. doi: 10.1097/ICL.0000000000000020. PMID 24508770